CLINICAL TRIAL: NCT04577222
Title: The Ability of Adipose Flap Over the NVB to Improve Sexual and Urinary Function Following Radical Prostatectomy; a Randomized Control Trial
Brief Title: The Ability of Adipose Flap Over the NVB to Improve Sexual and Urinary Function Following Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, golan shay, Doctor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 212-18
Record Dates: First submitted 2018-07-30; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer; Erectile Dysfunction; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose Flap (Experimental): Covering neurovascular bundle with fat
  Interventions: Procedure: Technical modification during radical prostatectomy
- Control (No Intervention): No adipose flap

INTERVENTIONS:
Procedure: Technical modification during radical prostatectomy — Covering the NVB with fat
  Arms: Adipose Flap

SUMMARY:
Despite technological advances, incontinence and impotence remain significant side effects of radical prostatectomy (RP). Strategies have been developed to reduce the injury to the erection nerves (i.e. neurovascular bundle - NVB)during surgery to further improve functional outcomes after RP. Adipose tissue is known for its stabilizing and even healing potential. These features include reducing the inflammatory process and improving blood supply to an injured nerve. We hypothesized that covering the NVB with periprostatic fat during surgery may potentially improve neural recovery and enhance functional recovery after RP. We sought to examine our hypothesis in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 years and older.
2. Patients diagnosed with prostate cancer.
3. Patients should be potent (IIEF erectile function domain score of 26 and above) and have a sexual partner.
4. Patients scheduled for Radical Prostatectomy with NVB preservation (at least unilateral).

Exclusion Criteria:

Patients who did not undergo NVB preservation or technical inability to create flap

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Erectile function | Change from Baseline IIEF score at 12 months
  IIEF erectile function score

SECONDARY OUTCOMES:
Continence status | Change from Baseline King's score at 12 months
  King's Health Questionnaire score

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel